CLINICAL TRIAL: NCT01421953
Title: Assessment of Four-dimensional (4D) 18F-fluoro-deoxy-glucose (FDG) Positron Emission Tomography and Computed Tomography System (PET-CT) in Radiotherapy for Non Small Cell Lung Cancers (NSCLC)
Brief Title: Assessment of 4D 18F-FDG PET-CT in Radiotherapy for Non Small Cell Lung Cancers
Acronym: PULMOTEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CHUBX 2011/01
Record Dates: First submitted 2011-08-11; First posted 2011-08-23 (Estimated); Last update posted 2014-10-23 (Estimated); Status verified 2014-10

CONDITIONS: Lung Cancer; Non-small-cell Lung Carcinoma
Keywords: Positron Emission Tomography; Computed Tomography; Lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Patients (Experimental)
  Interventions: Device: CT-simulation and 4D PET-CT

INTERVENTIONS:
Device: CT-simulation and 4D PET-CT — Patients will do a CT-simulation and 4D PET-CT in radiotherapy treatment position. The target volumes and the dosimetries obtained with both modalities will be compared.

SUMMARY:
Computed tomography (CT) images, used for radiotherapy planning, are often caught out in lung target volumes delineation because of their inability to differentiate between neoplasia, inflammation and atelectasia. Positron Emission Tomography (PET) is a new functional imaging modality and is currently used in the diagnosis and the staging of lung cancers. The aim of this study is to evaluate the impact of 4D 18F-FDG-PET-CT on radiotherapy planning for lung cancers.

DETAILED DESCRIPTION:
Many PET studies have been interested in lung radiotherapy volumes definition, however lacking any standardisation. Effectively, the use of PET images is difficult because of the poor image quality resulting from noise and partial volume effects induced blurring. Moreover, due to the long duration of PET acquisitions, respiratory motions are inevitable and result in artifacts in the PET images affecting the volumes and contrast of the tumour: tumours may appear larger while their activity can be lower. To overcome these limitations, we propose to use a 4D PET-CT, ie a PET-CT acquisition system synchronized with respiration in order to compare CT-simulation target volumes and PET target volumes after application of different approaches for partial volume effect correction, respiratory motion correction and automatic segmentation method of functional volumes. For this purpose, patients with a non small cell lung cancer and having to be treated with radiotherapy or radio-chemotherapy underwent CT-simulation and 4D PET-CT in radiotherapy treatment position. The target volumes and the dosimetries obtained with both modalities were compared.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18 years old
* patients with unresectable non small cell lung cancer having to be treated with radiotherapy or radio-chemotherapy

Exclusion Criteria:

* neo-adjuvant treatment
* patient treated previously with thoracic radiation
* patient unable to support 4D PET-CT
* pregnant or breast-feeding woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2011-08; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Quantitative and qualitative differences between CT-simulation and 4D PET-CT volumes | between day 7 and day 21 after inclusion
  Quantitative and qualitative differences between the radiotherapy target volumes obtained from CT-simulation and from 4D-PET-CT.
  The quantitative difference is expressed as a percentage of the total volume defined on CT simulation.
  The qualitative difference is defined as the volumes defined only on CT-simulation or only on 4D-PET-CT, expressed as a percentage of the total volume defined on CT-simulation.

SECONDARY OUTCOMES:
Dosimetrics differences between the dosimetries obtained from CT-simulation or from 4D-PET-CT. | between day 7 and day 21 after inclusion
Search of predictive criteria (histology, tumour localization, TNM staging) for 4D-PET-CT impact on the radiotherapy target volumes and on the dosimetries. | between day 7 and day 21 after inclusion

CONTACTS AND LOCATIONS:
Overall Officials: Philippe FERNANDEZ, Pr, Principal Investigator — University Hospital, Bordeaux, France
Locations (1):
- CHU Bordeaux - hôpital Pellegrin, Bordeaux, France